CLINICAL TRIAL: NCT03441997
Title: The Altered Immune Response to Exercise in Patients With Fibromyalgia Before and After a Mind-body Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00141263
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Fibromyalgia
Keywords: exercise; low intensity exercise; pain; fatigue; sleep problems
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain; Fatigue; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full mind-body exercises (Experimental): Participants will be trained to perform a type of mind-body exercise that involves low intensity exercise and body movements similar to Tai Chi. Participants will be asked to exercise 2 times per day for 8 weeks.
  Interventions: Other: Mind-body exercise
- Light mobility exercises: Control Group (Active Comparator): The Light mobility exercises group will perform a similar exercise as the experimental group. However without a few components. Participants will be asked to exercise two times per day for 8 weeks.
  Interventions: Other: Light mobility exercises
- Healthy Controls (No Intervention): Healthy females will be asked to make one visit to complete aerobic exercise test, questionnaires, and provide blood samples.

INTERVENTIONS:
Other: Mind-body exercise — Exercise program.
  Arms: Full mind-body exercises
Other: Light mobility exercises — Modified mind-body program.
  Arms: Light mobility exercises: Control Group

SUMMARY:
The purpose of this study is to compare two different exercise programs to see if there are differences after exercise in fibromyalgia (FM) symptoms and responses from the immune system.

ELIGIBILITY:
Inclusion Criteria for FM Patients:

* Patients with a diagnosis of FM
* Clearance from patient's physician to participate in a clinical trial
* Not participating or willing to discontinue FM treatment with trans-cutaneous electrical nerve stimulation, biofeedback, tender-point injections, acupuncture, Yoga, and Tai Chi.

Exclusion Criteria for all Participants:

* Diagnosis of severe psychiatric illness
* Abuse of alcohol, benzodiazepines, or other drugs
* Active cardiovascular, pulmonary, hepatic, renal, gastrointestinal, or autoimmune disease (except Hashimoto's or Graves' disease that has been stable for 3 months before screening)
* Current systemic infection
* Active cancer (except basal cell carcinoma);
* Unstable endocrine disease
* Severe sleep apnea
* Prostate enlargement or other genitourinary disorder (male patients)
* Pregnancy or breastfeeding

Inclusion Criteria for Healthy Controls:

* Female
* No apparent medical condition that will interfere with participation in the study
* Not on any medication that will interfere with participation in this study

Exclusion Criteria for Healthy Controls:

* Medical or surgical conditions including medication that preclude participation in the study
* Presence of motor or neuromuscular deficits that may preclude participating in fatigue exercise

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-17 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in anti-inflammatory cytokine (IL-6, IL-8, and IL-10) | At three time points: before exercise, at the maximum exertion, and 30 minutes after maximum exertion. This procedure will be conducted at baseline and after 8 weeks of qigong/sham-qigong practice.
  Changes will be measured during a bout of exhaustive exercise using a recumbent bicycle machine

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | At two time points: at baseline, and after 8 weeks of qigong/Sham-qigong intervention
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSIQ), which was designed to differentiate between good and poor sleepers. The PSIQ covers subjective sleep quality, sleep latency, sleep disturbances, sleep duration, daytime dysfunction and use of sleep medications. It consists of 19 self-rated questions. The PSIQ has been vastly employed in clinical trials, and it has been reported to be reliable and valid
Change in Pressure Pain Threshold (PPT) | At two time points: at baseline, and after 8 weeks of qigong/Sham-qigong intervention
  Pressure pain threshold is defined as the minimum force applied which induces pain. Mechanical pressure, determined as a kilogram (kg) per 1 cm2 of skin on the sensitive areas, is applied by a Fisher's hand dolorimeter. The examiner places the rubber tip on the examination site and gradually increases the pressure at a rate of approximately 1 kg per second. Subjects are instructed to say ''yes'' when the sensation of pressure causes pain and the pain pressure threshold is recorded. Pain threshold is measured in the 18 points specified by the American College of Rheumatology.
Change in Fibromyalgia Impact Questionnaire (FIQR) | At two time points: at baseline, and after 8 weeks of qigong/Sham-qigong intervention
  This questionnaire can capture the total spectrum of issues related to FM and the patient's response to therapies. It is one of the most used instrument in trials involving subjects with FM. Also, it has been proven to show consistent response to clinical changes
Change in Quality of Life evaluated by the Quality of Life Scale (QOLS) | At two time points: at baseline, and after 8 weeks of qigong/Sham-qigong intervention
  This scale is one of the most used instrument to measure quality of life in patients with chronic disease. The QOLS is a 15-item questionnaire that accesses five conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation. This scale has been shown to be reliable and validated by previous studies

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Sarmento CVM, Moon S, Pfeifer T, Smirnova IV, Colgrove Y, Lai SM, Liu W. The therapeutic efficacy of Qigong exercise on the main symptoms of fibromyalgia: A pilot randomized clinical trial. Integr Med Res. 2020 Dec;9(4):100416. doi: 10.1016/j.imr.2020.100416. Epub 2020 Apr 25. PMID 32455108